CLINICAL TRIAL: NCT06483958
Title: Palliative Care Protocol for Adult Patients at High Risk of Death in Critical Care Units: A Multicentric Stepped Wedge Cluster Randomised Trial
Brief Title: Palliative Care Protocol for Adult Patients Hospitalized in Critical Care Units.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OAIC 1315/22
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-01

CONDITIONS: End of Life Care; Critical Illness; Palliative Care
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Palliative care protocol
  Interventions: Behavioral: palliative care protocol
- Standard care (No Intervention): None intervention

INTERVENTIONS:
Behavioral: palliative care protocol — 1. Symptom management
  2. Respect for patient and family autonomy.
  3. Respectful management of clinical information.
  4. Provision of holistic care and support.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to determine the effectiveness of a palliative care protocol in improving the quality of care of adult patients at high risk of dying hospitalized in the critical care unit.

Assessing symptom burden (dyspnea, pain and/or anxiety/agitation) until death or day 5 (whichever comes first)

Researchers will compare the impact of the palliative care protocol with standard care to see if it improves the quality of care.

Participants will:

1. Symptom management.
2. Respect for the autonomy of the patient and his/her family environment.
3. Respectful management of clinical information.
4. Provision of holistic care and support.

DETAILED DESCRIPTION:
We designed a stepped wedge cluster randomized trial The study is implementation in 5 Chilean hospitals, admitting 248 patients.

Pre-intervention (control): The practices of each ICU will be maintained, until the moment that according to randomization corresponds the beginning of the intervention, in each center.

Post-intervention: Palliative care protocol to improve the quality of care

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* Hospitalization in critical care unit for more than 48 hrs.
* Medical indication of therapeutic effort limitation, defined as: a) Non-initiation or withdrawal of life support therapies: invasive mechanical ventilation, vasoactive drugs, cardiopulmonary resuscitation, renal replacement therapy.

Exclusion Criteria:

* Severe communication disorder and cultural language limitation (language other than Spanish).
* Absence of legal representative and/or caregiver.
* Brain dead patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Burden of symptoms present in the last 24 hours prior to death (or end of follow-up). | From recruitment until death or day 5 of follow up
  The percentage of patients with at least one episode of pain, dyspnea, agitation, or anxiety

SECONDARY OUTCOMES:
Family satisfaction | Up to 4 week after death or hospital discharge
  Family satisfaction in relatives of adult patients at high risk of death.

CONTACTS AND LOCATIONS:
Locations (1):
- Verónica Rojas, Santiago, Me, Chile

IPD SHARING:
Plan to Share IPD: No